CLINICAL TRIAL: NCT00598715
Title: Randomized Trial of Paclitaxel- vs Sirolimus-eluting Stents for Treatment of Coronary Restenosis in Sirolimus-eluting Stents
Brief Title: Efficacy Study of Two Different Strategies for Restenosis in Sirolimus-Eluting Stents
Acronym: DESIRE-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Albert Schomig, Deutsches Herzzentrum Muenchen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GE IDE No. S02407
Record Dates: First submitted 2008-01-10; First posted 2008-01-22 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2009-09

CONDITIONS: Coronary Artery Disease
Keywords: In-stent restenosis; In-DES-restenosis; paclitaxel; sirolimus
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Same drug (Experimental): sirolimus-eluting stent will be implanted for restenosis after previous the implantation of a sirolimus-eluting stent
  Interventions: Device: Sirolimus eluting stent
- Different drug (Active Comparator): paclitaxel eluting stent will be implanted for restenosis after previous the implantation of a sirolimus-eluting stent
  Interventions: Device: Paclitaxel-eluting stent

INTERVENTIONS:
Device: Sirolimus eluting stent — Sirolimus-eluting stent will be implanted
  Other Names: Cypher
  Arms: Same drug
Device: Paclitaxel-eluting stent — Paclitaxel-eluting stent will be implanted
  Other Names: Taxus
  Arms: Different drug

SUMMARY:
For lesions which develop restenosis after a drug-eluting stent, it is not known which the right strategy to use is, implantation of the same type of DES as the initial one or a DES with a different drug.

DETAILED DESCRIPTION:
Treatment of in-stent restenosis after implantation of a DES has poorly been studied. Although there are no data, it may be assumed that certain lesions might be resistant to a given drug and in need of a different DES. Thus, for lesions which develop restenosis after a DES, it is not known which the right strategy to use is, implantation of the same type of DES as the initial one or a DES with a different drug. This prospective, randomized trial will compare the anti-restenotic efficacy of PES or SES in patients with restenosis after initial implantation of a SES

ELIGIBILITY:
Inclusion Criteria:

* Patients older than age 18 with ischemic symptoms or evidence of myocardial ischemia in the presence of > 50% re- stenosis after prior implantation of Sirolimus eluting stents in native coronary vessels
* Written, informed consent by the patient or her/his legally-authorized representative for participation in the study
* In women with childbearing potential a negative pregnancy test is mandatory

Exclusion Criteria:

* Cardiogenic shock
* Acute myocardial infarction within the first 48 hours from symptom onset.
* Target lesion located in the left main trunk or bypass graft.
* Malignancies or other comorbid conditions (for example severe liver, renal and pancreatic disease) with life expectancy less than 12 months or that may result in protocol non-compliance.
* Allergy to antiplatelet therapy, sirolimus, paclitaxel, stainless steel.
* Pregnancy (present, suspected or planned) or positive pregnancy test.
* Previous enrollment in this trial.
* Patient's inability to fully comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2007-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Late luminal loss at follow-up angiography | 6-8 months

SECONDARY OUTCOMES:
Need of target lesion revascularization. | 12 months
Combined incidence of death or myocardial infarction. | 12 months
Incidence of stent thrombosis. | 12 months
Incidence of binary restenosis at follow-up angiography | 6-8 months

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Kastrati, MD, Principal Investigator — Deutsches Herzzentrum Muenchen; Julinda Mehilli, MD, Study Director — Deutsches Herzzentrum Muenchen
Locations (2):
- Germany (2):
  - Deutsches Herzzentrum Muenchen, Munich
  - 1. Medizinische Klinik, Klinikum rechts der Isar, Munich

REFERENCES:
- [Background] Kastrati A, Mehilli J, von Beckerath N, Dibra A, Hausleiter J, Pache J, Schuhlen H, Schmitt C, Dirschinger J, Schomig A; ISAR-DESIRE Study Investigators. Sirolimus-eluting stent or paclitaxel-eluting stent vs balloon angioplasty for prevention of recurrences in patients with coronary in-stent restenosis: a randomized controlled trial. JAMA. 2005 Jan 12;293(2):165-71. doi: 10.1001/jama.293.2.165. PMID 15644543
- [Result] Mehilli J, Byrne RA, Tiroch K, Pinieck S, Schulz S, Kufner S, Massberg S, Laugwitz KL, Schomig A, Kastrati A; ISAR-DESIRE 2 Investigators. Randomized trial of paclitaxel- versus sirolimus-eluting stents for treatment of coronary restenosis in sirolimus-eluting stents: the ISAR-DESIRE 2 (Intracoronary Stenting and Angiographic Results: Drug Eluting Stents for In-Stent Restenosis 2) study. J Am Coll Cardiol. 2010 Jun 15;55(24):2710-6. doi: 10.1016/j.jacc.2010.02.009. Epub 2010 Mar 11. PMID 20226618
- [Derived] Kufner S, Byrne RA, de Waha A, Schulz S, Joner M, Laugwitz KL, Kastrati A; Intracoronary Stenting and Angiographic Results: Drug Eluting Stents for In-Stent Restenosis 2, (ISAR-DESIRE 2) Investigators. Sirolimus-eluting versus paclitaxel-eluting stents in diabetic and non-diabetic patients within sirolimus-eluting stent restenosis: results from the ISAR-DESIRE 2 trial. Cardiovasc Revasc Med. 2014 Mar;15(2):69-75. doi: 10.1016/j.carrev.2014.02.001. Epub 2014 Feb 15. PMID 24684757